CLINICAL TRIAL: NCT02050464
Title: Virtual Physiological Human (VPH) Dementia Research Enabled by IT - Prospective Cohort Kuopio
Brief Title: Computational Tools for Early Diagnosis of Memory Disorders
Acronym: ProsKuopio
Status: Completed | Type: Observational
Sponsor: University of Eastern Finland (Other)
Collaborators: University of Sheffield (Other); VTT Technical Research Centre of Finland (Other); Klinik Hirslanden, Zurich (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Hilkka Soininen, Hilkka Soininen, Professor, MD, PhD, University of Eastern Finland
Other Study IDs: 207094
Record Dates: First submitted 2014-01-15; First posted 2014-01-30 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Alzheimer Disease; Frontotemporal Dementia; Dementia, Vascular; Mild Cognitive Impairment
Keywords: Alzheimer Disease; Frontotemporal Dementia; Dementia, Vascular; Mild Cognitive Impairment; Diagnosis; Risk factors; Biomarkers; AD; FTD; VAD; MCI
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia; Dementia, Vascular; Cognitive Dysfunction; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, white cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Healthy controls: Healthy controls
- Alzheimer's disease: Patients with mild Alzheimer's disease
- Vascular dementia: Patients with vascular dementia
- Fronto-temporal dementia: Patients with fronto-temporal dementia
- Mild cognitive impairment: Patients with mild cognitive impairment

SUMMARY:
The Virtual Physiological Human: DementiA Research Enabled by IT (VPH-DARE@IT) is a four-year IT-project funded through the European Union (EU). The project consortium involves a total of 21 universities and industrial partners from 10 European countries. The project delivers the first patient-specific predictive models for early differential diagnosis of dementia and their evolution. An integrated clinical decision support platform will be validated / tested by access to a dozen databases of international cross-sectional and longitudinal studies. As a part of the VPH-DARE@IT project, a new prospective cohort will be collected in Kuopio. This prospective cohort will be used to test further the modeling approaches and tools developed by using the retrospective databases.

DETAILED DESCRIPTION:
The Virtual Physiological Human: DementiA Research Enabled by IT (VPH-DARE@IT) is a four-year IT-project funded through the European Union (EU). The project will develop multiscale models of the ageing brain in order to account simultaneously for the patient-specific biochemical, metabolic and biomechanical brain substrate, as well as for genetic, clinical, demographic and lifestyle determinants. An integrated clinical decision support platform will be validated and tested by access to a dozen databases of international cross-sectional and longitudinal studies.

Modeling approaches developed by using the retrospective databases will be tested using a new prospective cohort that will be collected in Kuopio as a part of the VPH-DARE@IT project. The study population at university of Eastern Finland (UEF) will be a total of 120 subjects: 20 healthy controls (HC), 20 mild to moderate Alzheimer's disease (AD) patients, 20 vascular dementia (VAD) patients, 20 fronto-temporal dementia (FTD) patients and 40 subjects with mild cognitive impairment (MCI). This study is referred as VPH-DARE@IT Prospective study in Kuopio or "ProsKuopio".

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for subjects with dementia (AD, VAD, FTD) - The inclusion criteria will be based on international research criteria:

* Diagnosis of probable AD according to National Institute of Neurological and Communicative Disorders and Stroke Alzheimer's (NINCDS-ADRDA) criteria (McKhann et al.1984) and diagnosis of prodromal AD according to Dubois et al., 2007 criteria
* Diagnosis of FTD according to the clinical diagnostic criteria of Neary et al., 1998
* Diagnosis of VAD according to diagnostic criteria for research studies by the NINDSAIREN International Workshop (Román et al., 1993)

Inclusion criteria for subjects with MCI

* Referral because of cognitive impairments
* Diagnosis criteria for amnestic and nonamnestic MCI (Petersen, 2004, Petersen and Morris, 2005)

Inclusion criteria for control subjects

* Mini-mental state examination (MMSE) score above or equal to 27
* Overall score on the Clinical Dementia Rating (CDR) scale of 0

Exclusion Criteria:

Exclusion criteria for all subjects

* Other causes of dementia
* Obvious brain, systemic or psychiatric disorders that could potentially affect cognitive functions such as stroke, severe depression, or endocrine disorders

Exclusion criteria for control subjects and subjects with MCI

- Diagnosis of dementia according to DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, 4th Edition) criteria at baseline

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Control subjects with normal cognition
  The Alzheimer's disease, Fronto-temporal dementia, Vascular dementia, and Mild Cognitive Impairment will be recruited during their visit in the Neurological clinic at the Kuopio University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2013-12; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity and accuracy of models for diagnosis of memory disorders | during a single visit, i.e., day 1 and for one study group (MCI) after 18 month follow-up
  The models developed the VPH-DARE project will be tested in this prospective cohort. Sensitivity, specificity and accuracy of the model will be tested in differential diagnosis between the study groups as well as the accuracy of prediction cognitive decline as measured by neuropsychological test battery in the MCI group.

CONTACTS AND LOCATIONS:
Overall Officials: Hilkka Soininen, Professor, Principal Investigator — University of Eastern Finland
Locations (3):
- Finland (3):
  - Department of Neurology and Brain Research Unit, Institute of Clinical Medicine, University of Eastern Finland, Kuopio
  - Kuopio University Hospital, Kuopio
  - VTT Technical Research Centre of Finland, Tampere

REFERENCES:
- See also: Click here for more information about VPH-DARE@IT project — http://www.vph-dare.eu